CLINICAL TRIAL: NCT04816539
Title: Comparison of the TOFscan and the TetraGraph During Recovery of Neuromuscular Function : a Pilot Study
Brief Title: Comparison of the TOFscan and the TetraGraph During Recovery of Neuromuscular Function
Acronym: DECURAR-EMG
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-A03054-35
Record Dates: First submitted 2021-03-23; First posted 2021-03-25 (Actual); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: Neuromuscular Blockade

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: TetraGraph — Use of two monitoring devices of neuromuscular function during surgery

SUMMARY:
Assess the values of train-of-four ratios with the TetraGraph and thoses obtained with the TOFscan during recovery of neuromusculat function in surgical patients who have been administred rocuronium.

Primary outcome : value of TOFratio with the TetraGraph when TOFratio of TOFscan is greater than or equal to 90% Pilot study : no hypothesis

ELIGIBILITY:
Inclusion Criteria:

* age greater than or equal to 18 years old
* patients willing to participate and provide an informed consent
* elective surgical procedures, without emergency, administration of rocuronium for neuromuscular blockade, and recovery of complete neuromuscular function at the end of the surgery

Exclusion Criteria:

* patients with unilateral disorders, such as stroke, carpal tunnel syndrome, broken wrist with nerve damage, Dupuytren contracture, or similar wrist injury
* patients with systemic neuromuscular diseases such as myasthenia gravis
* renal insufficiency or renal failure
* significant liver disease
* patients having surgery that would involve prepping the arm into the sterile field
* allergy to rocuronium

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing an electrive surgical procedure with non emergency and that requires use of Rocuronium, and willing to participate and provide an informed consent
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-04-15 (Estimated); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
Train-of-four ratios | baseline (J0)
  Value of TOFratio with TetraGraph when TOFratio with TOFscan is greater than or equal to 90% (first value of three greater than or equal to 90%)

SECONDARY OUTCOMES:
Train-of-four ratios | baseline (J0)
  Value of TOFratio with TetraGraph when TOFratio with TOFscan is greater than or equal to 10%, 20%, 30%, 40%, 50%, 60%, 70%, 80% and eventually 100%
Train-of-four ratios | baseline (J0)
  Value of TOFratio with TOFscan when TOFratio with TetraGraph is greater than or equal to 10%, 20%, 30%, 40%, 50%, 60%, 70%, 80% and eventually 100%
Train-of-four count | baseline (J0)
  Time to recover one, two, three and four responses from TOFcount with TOFscan and TetraGraph

CONTACTS AND LOCATIONS:
Overall Officials: Claude Meistelman, Principal Investigator — CHU NANCY
Locations (1):
- Chu Nancy, Vandœuvre-lès-Nancy, France